CLINICAL TRIAL: NCT04097444
Title: Quadruplet 1st Line Treatment of CAPOXIRI Plus Bevacizumab Versus FOLFOXIRI Plus Bevacizumab for mCRC, Multicenter Randomised Phase II Study (QUATTRO-II)
Brief Title: CAPOXIRI+Bevacizumab vs. FOLFOXIRI+Bevacizumab for mCRC
Acronym: QUATTRO-II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QUATTRO-II
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; bevacizumab; CAPOXIRI; FOLFOXIRI
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Fluorouracil; Leucovorin; Irinotecan; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Step 1 (CAPOXIRI+ BEV) (Experimental): Induction therapy is followed by the maintenance therapy.
  [Induction treatment: CAPOXIRI+BEV] Administered for 6 cycles (a maximum of 8 cycles). BEV: 7.5mg/kg (d.i.v.) oxaliplatin (OX): 100/130 mg/sq.m (d.i.v.) irinotecan (IRI):150/180/200mg/sq.m (d.i.v.) CAP 1,600 mg/sq.m /day (p.o. day1-15) Administered every 3 weeks. OX/IRI dose is applied according to the progress of Step 1.
  [Maintenance treatment: 5-fluorouracil (FU)/Levofolinate calcium (LV)+BEV or CAP+BEV] The following 5-FU/LV+BEV therapy will be repeated in 2-week cycles, or the following CAP+BEV therapy will be repeated in 3-week cycles (Physician's choice). No change in treatment regimen will be permitted after the selection of maintenance therapy (5-FU/LV+BEV or CAP+ BEV).
  5-FU/LV+BEV: BEV:5mg/kg (d.i.v.) l-LV:200mg/sq.m (d.i.v.) 5-FU:3,200mg/sq.m (c.i.v.) Administered every 2 weeks.
  CAP+BEV: BEV: 7.5mg/kg (d.i.v.) CAP 1,600 mg/sq.m /day (po. day1-15) Administered every 3 weeks.
  Interventions: Biological: Bevacizumab; Drug: Irinotecan hydrochloride; Drug: Oxaliplatin; Drug: Capecitabine
- Step 2 Arm A (FOLFOXIRI+ BEV) (Experimental): Induction therapy is followed by the maintenance therapy.
  [Induction treatment: FOLFOXIRI+BEV] Administered for 8 cycles (a maximum of 12 cycles). BEV: 5mg/kg (d.i.v.) OX: 85 mg/sq.m (d.i.v.) IRI:165mg/sq.m (d.i.v.) LV:200mg/sq.m (d.i.v.) 5-FU:3,200mg/sq.m (c.i.v.) Administered every 2 weeks.
  [Maintenance treatment: 5-FU/LV+BEV or CAP+BEV] The following 5-FU/LV+BEV therapy will be repeated in 2-week cycles, or the following CAP+BEV therapy will be repeated in 3-week cycles (Physician's choice). No change in treatment regimen will be permitted after the selection of maintenance therapy (5-FU/LV+BEV or CAP+ BEV).
  5-FU/LV+BEV: BEV:5mg/kg (d.i.v.) LV:200mg/sq.m (d.i.v.) 5-FU:3,200mg/sq.m (c.i.v.) Administered every 2 weeks.
  CAP+BEV: BEV: 7.5mg/kg (d.i.v.) CAP 1,600 mg/sq.m /day (po. Day1-15) Administered every 3 weeks.
  Interventions: Biological: Bevacizumab; Drug: 5-fluorouracil; Drug: Leucovorin calcium; Drug: Irinotecan hydrochloride; Drug: Oxaliplatin
- Step 2 Arm B (CAPOXIRI+ BEV) (Experimental): Induction therapy is followed by the maintenance therapy.
  [Induction treatment: CAPOXIRI+BEV] Administered for 6 cycles (a maximum of 8 cycles). BEV: 7.5mg/kg (d.i.v.) OX: 100/130 mg/sq.m (d.i.v.) IRI:150/180/200mg/sq.m (d.i.v.) CAP 1,600 mg/sq.m /day (p.o. day1-15) Administered every 3 weeks. Regarding to OX/IRI dose, RD will be confirmed at Step 1.
  [Maintenance treatment: 5-FU/LV+BEV or CAP+BEV] The following 5-FU/LV+BEV therapy will be repeated in 2-week cycles, or the following CAP+BEV therapy will be repeated in 3-week cycles (Physician's choice). No change in treatment regimen will be permitted after the selection of maintenance therapy (5-FU/LV+BEV or CAP+ BEV).
  5-FU/LV+BEV: BEV:5mg/kg (d.i.v.) l-LV:200mg/sq.m (d.i.v.) 5-FU:3,200mg/sq.m (c.i.v.) Administered every 2 weeks.
  CAP+BEV: BEV: 7.5mg/kg (d.i.v.) CAP 1,600 mg/sq.m /day (po. day1-15) Administered every 3 weeks.
  Interventions: Biological: Bevacizumab; Drug: Irinotecan hydrochloride; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: BEV
Drug: 5-fluorouracil — Given IV
  Other Names: 5-FU
  Arms: Step 2 Arm A (FOLFOXIRI+ BEV)
Drug: Leucovorin calcium — Given IV
  Other Names: LV
  Arms: Step 2 Arm A (FOLFOXIRI+ BEV)
Drug: Irinotecan hydrochloride — Given IV
  Other Names: IRI
Drug: Oxaliplatin — Given IV
  Other Names: OX
Drug: Capecitabine — Given PO
  Other Names: CAP
  Arms: Step 1 (CAPOXIRI+ BEV); Step 2 Arm B (CAPOXIRI+ BEV)

SUMMARY:
The objective is to compare the efficacy and safety of CAPOXIRI+BEV therapy versus FOLFOXIRI+BEV therapy as first-line therapy in patients with metastatic colorectal cancer (mCRC).

DETAILED DESCRIPTION:
QUATTRO-II is an open-label, multicenter, randomised, phase II study to investigate the efficacy and safety of CAPOXIRI+BEV versus FOLFOXIRI+BEV in 1st line mCRC.

This study is composed two steps because of confirming of recommended dose (RD) for CAPOXIRI+BEV regimen.

1. Dose finding step (Step1): CAPOXIRI+BEV doses findings were planned by 3+3 cohort design, register up to maximum of 12 cases.
2. Randomised step (Step2): After confirmation of RD regarding CAPOXIRI+BEV, we will move to Step2 to compare the efficacy and safety between FOLFOXIRI+BEV and CAPOXIRI+BEV, register up to 65 cases.

ELIGIBILITY:
Inclusion Criteria:

1. Personal written informed consent is obtained after the study has been fully explained
2. Histologically confirmed colon or rectal adenocarcinoma

   *Excluding appendix cancer and anal canal cancer
3. Clinically unresectable
4. ≥20 years of age at enrollment
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1 (≥71 years of age: PS score of 0)
6. Measurable lesion according to RECIST ver. 1.1 criteria on contrast-enhanced chest, abdominal, or pelvic (trunk) CT (required within 28 days of enrollment)
7. No previous chemotherapy for colon or rectal cancer

   *Patients with confirmed relapse ≥24 weeks after completion of post-operative adjuvant chemotherapy can be enrolled
8. Ras/Braf mutation analysis at enrollment identifies Ras/Braf status as either the wild type or mutant type.
9. Vital organ functions meet the following criteria within 14 days before enrollment.

   If multiple test results are available in that period, the results closest to enrollment will be used. No blood transfusions or hematopoietic factor administration will be permitted within 2 weeks before the date on which measurements are taken.

   i. Neutrophil count: ≥1,500 /cu.mm

   ii. Platelet count: ≥10.0 × 104/cu.mm

   iii. Hemoglobin concentration: ≥9.0 g/dL

   iv. Total bilirubin: ≤1.5 times upper limit of normal (ULN)

   v. Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Alkaline phosphatase (ALP): ≤2.5 times ULN (≤5 times ULN for metastases to liver)

   vi. Serum creatinine: ≤1.5 times ULN, or creatinine clearance: ≥30 mL/min

   vii. Urine protein: ≤2+ (if ≥3+, urine protein/creatinine ratio: <2.0)
10. UGT1A1 polymorphism is wild type or single heterozygous type -

Exclusion Criteria:

1. Previous radiation therapy in which ≥20% bone marrow was exposed to the radiation field
2. Untreated brain metastases, spinal cord compression, or primary brain tumor
3. History of central nervous system (CNS) disease (excluding asymptomatic lacunar infarction)
4. Continuous systemic corticosteroid treatment is required
5. Oral or parenteral (such as low molecular weight heparin) anticoagulant dose is not consistently (≥14 days) controlled. (Oral anticoagulants: conditions at high risk for bleeding, such as prothrombin time (PT)-international normalized ratio (INR) ≥3, clinically significant active bleeding (within 14 days of enrollment))
6. Evidence of cardiovascular disease, cerebrovascular disorder (within 24 weeks), myocardial infarction (within 24 weeks), unstable angina pectoris, New York Heart Association (NYHA) classification ≥Grade II congestive heart failure, serious arrhythmias requiring drug therapy
7. Previous treatment with an investigational drug within 28 days prior to enrollment, or participation in a study of an unapproved drug
8. Any of the following comorbidities

   i. Uncontrolled hypertension

   ii. Uncontrolled diabetes mellitus

   iii. Uncontrolled diarrhea

   iv. Peripheral sensory neuropathy (≥Grade 1)

   v. Active peptic ulcer

   vi. Unhealed wound (except for suturing associated with implanted port placement)

   vii. Other clinically significant disease (such as interstitial pneumonia or renal impairment)
9. Major surgical procedure within 28 days prior to study treatment initiation (such as open chest, laparoscopy, thoracoscopic surgery, laparoscopic surgery), unless only colostomy is performed; open biopsy or suturing for major trauma within 14 days of study treatment initiation; or planned major surgical procedure during the study (open chest, laparoscopy) ("major surgical procedures" does not include central venous (CV) port insertion)
10. Physical defects of the upper gastrointestinal tract; malabsorption syndrome or difficulty taking oral medication
11. Pregnant, breastfeeding, positive pregnancy test (women who have menstruated in the last year will be tested), or women who are unwilling to use contraception; men who are unwilling to use contraception during the study
12. Active hepatitis B or C, or evidence of HIV infection
13. Previous chemotherapy for other malignancies (excluding hormone therapy for breast cancer)
14. Other active malignancies (synchronous malignancies, and asynchronous malignancies separated by a 5-year disease-free interval) (excluding malignancies that are expected to be completely cured, such as intramucosal carcinoma and carcinoma in situ)
15. Uncontrolled venous thromboembolism (unless clinically stable, asymptomatic, or appropriately treated with an anticoagulant)
16. Arterial thrombosis or arterial thromboembolism such as myocardial infarction, transient ischemic attack, or cerebrovascular attack in the last year prior to enrollment
17. Complications such as intestinal paralysis, intestinal obstruction, or gastrointestinal perforation, current or within 1 year prior to enrollment
18. Pleural effusion, ascites, or pericardial effusion requiring drainage
19. History of hypersensitivity to fluorouracil, levofolinate, oxaliplatin, irinotecan, bevacizumab and their excipients or Chinese hamster ovary cell proteins
20. History of adverse reactions to fluoropyrimidine drugs indicative of dihydropyrimidine dehydrogenase (DPD) deficiency
21. Systemic treatment required for, or evidence of, infections
22. Endoluminal stenting
23. Otherwise unsuitable for the study in the opinion of investigators -

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2019-10-11 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 18 months
  PFS by investigator-reported measurements according to CT image. PFS was calculated from the day of treatment start to the first observation of progression disease (PD) or death from any cause.PD was defined as Overall Response by RECIST criteria v1.1 according to CT image.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 36 months
Overall survival (OS) | Up to 36 months
Incidence of adverse events | Up to 36 months
  Adverse events were evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0. All adverse events was collected in duration from starting treatment to whichever shorter "after 30 days from withdrawal treatment" or "later treatment
Functional Assessment of Cancer Therapy (FACT) / Gynaecologic Oncology Group (GOG) Neurotoxicity 4 | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kato, M.D., Ph.D., Principal Investigator — Department of Surgery, National Hospital Organization Osaka National Hospital.; Akihito Tsuji, M.D., Ph.D., Principal Investigator — Department of Medical Oncology, Kagawa University Hospital.
Locations (1):
- Ac Medical Inc., Chuo Ku, Tokyo, Japan

REFERENCES:
- [Derived] Bando H, Kotani D, Satake H, Hamaguchi T, Shiozawa M, Kotaka M, Masuishi T, Yasui H, Kagawa Y, Komatsu Y, Oki E, Yamamoto Y, Kawakami H, Misumi T, Taniguchi H, Yamazaki K, Muro K, Yoshino T, Kato T, Tsuji A. QUATTRO-II randomized trial: CAPOXIRI+bevacizumab vs. FOLFOXIRI+bevacizumab as first-line treatment in patients with mCRC. Med. 2024 Sep 13;5(9):1164-1177.e3. doi: 10.1016/j.medj.2024.05.012. Epub 2024 Jun 19. PMID 38901425
- [Derived] Kotani D, Yoshino T, Kotaka M, Kawazoe A, Masuishi T, Taniguchi H, Yamazaki K, Yamanaka T, Oki E, Muro K, Komatsu Y, Bando H, Satake H, Kato T, Tsuji A. Combination therapy of capecitabine, irinotecan, oxaliplatin, and bevacizumab as a first-line treatment for metastatic colorectal cancer: Safety lead-in results from the QUATTRO-II study. Invest New Drugs. 2021 Dec;39(6):1649-1655. doi: 10.1007/s10637-021-01125-2. Epub 2021 May 21. PMID 34019214
- [Derived] Miyo M, Kato T, Yoshino T, Yamanaka T, Bando H, Satake H, Yamazaki K, Taniguchi H, Oki E, Kotaka M, Oba K, Miyata Y, Muro K, Komatsu Y, Baba H, Tsuji A. Protocol of the QUATTRO-II study: a multicenter randomized phase II study comparing CAPOXIRI plus bevacizumab with FOLFOXIRI plus bevacizumab as a first-line treatment in patients with metastatic colorectal cancer. BMC Cancer. 2020 Jul 23;20(1):687. doi: 10.1186/s12885-020-07186-5. PMID 32703200